CLINICAL TRIAL: NCT02923661
Title: Patient Satisfaction in Single Implant Mandibular Complete Overdentures Retained by CM LOC Versus Ball Attachment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Karim Fouda, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-09-205
Record Dates: First submitted 2016-10-02; First posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Edentulous; Dental Implant
Keywords: single implant
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CM LOC attachment group (Experimental): this group will receive CM LOC attachment and lower overdenture attached to it
  Interventions: Device: CM LOC
- Ball attachment (Active Comparator): this group will receive Ball attachment and lower overdenture attached to it
  Interventions: Device: ball attachment

INTERVENTIONS:
Device: CM LOC
  Other Names: Resin matrix
  Arms: CM LOC attachment group
Device: ball attachment
  Arms: Ball attachment

SUMMARY:
this study was conducted to clarify the effect of two different attachments on patient satisfaction and marginal bone loss. The primary and secondary objectives are to determine patient satisfaction and the marginal bone loss around implant when using CM LOC compared to conventional ball attachment. all the patients will receive a single median implant to which the denture will be loaded upon using the two different attachment systems

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous male or female patients between the ages of 50 to 69.
* No contraindications for implantation.
* Each patient has to perform both a random blood sugar and Glycosylated Hemoglobin analysis. Patients with a Glycosylated hemoglobin test HbA1c up to 8% and a normal blood sugar level (79 to 110) or controlled diabetic patients (90-130 fasting according to American Association of Diabetes) will be included.
* Sufficient bone width (≥ 6 mm) in the anterior region to place an implant. It could be either normally present or achieved by bone plateauing. This will be confirmed by cone beam computed tomographic (CBCT) scans.
* Residual bone height ranging from 11-20 mm with the lowest vertical height in the midline of the mandible not less than 13 mm (Class II or III according to McGarry et al.22This will be confirmed by the CBCT.
* Patients seeking to install a single symphyseal implant and for whom new dentures will be constructed.
* Patients, who are dissatisfied with the retention and stability of their technically satisfactory dentures.
* Patients, who already have existing maxillary and mandibular complete dentures, and after examination of the mandibular dentures, it is found that there are technical problems with regard to denture design and/or occlusion; then new maxillary and mandibular dentures will be fabricated
* All patients should have adapted to their dentures for at least six weeks before being included in the trial.
* Patients providing written informed consents to participate in the trial and this will be done before the scheduled date for implant installation.

Exclusion Criteria:

* Patients with a systemic or local contra-indication for implant placement.
* Satisfied patients with the retention of their mandibular denture as well as unsatisfied patients with their maxillary denture.
* Patient with a mandibular denture height less than 6 mm between the base of the denture and the incisal edge of the central incisors (as measured by a caliper) or with 12 mm crown height space as measured by a ruler from the incisal edge till the crest of the ridge. This will be done from a putty index of the diagnostic set up.
* Incompliant and not cooperative patients.
* Patients smoking more than 10 cigarettes per day

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | 1 year
  patient satisfaction will be measured using a questionnaire

SECONDARY OUTCOMES:
Marginal bone loss | 1 year
  Marginal bone loss will be measured using paralleling radiography

CONTACTS AND LOCATIONS:
Overall Officials: Karim M. Fouda, Master, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided